CLINICAL TRIAL: NCT02097056
Title: Safety and Efficacy of Donepezil HCl 23 mg in Patients With Moderate to Severe Alzheimer's Disease
Acronym: SAVE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eisai Korea Inc. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ART-M082-401
Record Dates: First submitted 2014-03-24; First posted 2014-03-26 (Estimated); Results first posted 2016-06-27 (Estimated); Last update posted 2016-06-27 (Estimated); Status verified 2016-05

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Donepezil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- donepezil HCl 23 mg (Experimental): Donepezil HCl 23 mg once daily, just before bed, for 24 weeks
  Interventions: Drug: Donepezil HCL

INTERVENTIONS:
Drug: Donepezil HCL — Donepezil HCl 23 mg once daily, just before bed, for 24 weeks

SUMMARY:
This is a multi-center, open-label, single-arm, prospective, phase IV trial, evaluating safety and efficacy of donepezil hydrochloride in patients with moderate to severe Alzheimer's disease.

DETAILED DESCRIPTION:
This study consisted of pre-treatment and treatment phase. Pre-treatment phase was approximately 4 weeks including the screening and baseline process. In treatment phase, about 190 subjects received Donepezil HCl 23 mg once daily for 24 weeks.

ELIGIBILITY:
Inclusion Criteria

1. Male or female aged 45 to 90 years
2. Patients have eligible conditions of dementia diagnosis listed in DSM-IV
3. Diagnosed as a probable Alzheimer's Disease patient according to NINCDS-ADRDA criteria
4. At the timing of screening, MMSE less than or equal to 20 AND CDR greater than or equal to 2 OR GDS greater than or equal to 4
5. Patients, who have been taking stable donepezil 10 mg for 3 months or longer before the start of the study (screening visit), are evaluated as eligible to take donepezil 23 mg by investigator
6. Patients who have not received any other medications for AD such as AChE inhibitors at least for 3 months prior to the screening visit excluding donepezil hydrochloride (However, concomitant use of memantine is allowed if taken at stable dose that are less than or equal to the approved dose range for at least 3 months prior to screening)
7. Medicines for cerebral activation such as Gingko Biloba is allowed to be taken if the patient has received it as stable dose for 3 months prior to the screening visit

Exclusion Criteria

1. Patients who have been participated in any other clinical trial 3 months prior to the screening visit
2. Patients who are having any severe psychiatric disorder or schizophrenia
3. Patients who are having a neurological disorder other than AD which affect the subject's cognition or ability to assess the cognition

Ages: 45 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 171 (Actual)
Dates: Start 2014-02; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (13):
- South Korea (13):
  - Ansan, Gyeonggi-do
  - Buchoen, Gyeonggi-do
  - Seongnam-si, Gyeonggi-do
  - Jinju, Gyeongsangnam-do
  - Iksan, Jeollabuk-do
  - Hwasun, Jeollanam-do
  - Busan, Korea, Republic of
  - Daegu, Korea, Republic of
  - Daejeon, Korea, Republic of
  - Incheon, Korea, Republic of
  - Jeju City, Korea, Republic of
  - Seoul, Korea, Republic of
  - Chungju, North Chungcheong

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Out of the 171 participants enrolled into the study, 1 was not treated resulting in 170 participants in the safety population.
Groups:
- Donepezil Hydrochloride: Donepezil hydrochloride (HCl) at 23 mg was administered once daily, just before bed, for 24 weeks.
Period: Overall Study
Arm/Group | Donepezil Hydrochloride
Started | 171
ParticipantsTreated | 170
Completed | 113
Not Completed | 58
Not completed — Protocol Violation | 2
Not completed — Withdrawal by Subject | 15
Not completed — Lost to Follow-up | 2
Not completed — Adverse Event | 37
Not completed — Other | 2

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who received at least one dose of study treatment and had at least one postbaseline safety assessment.
Arm/Group | Donepezil Hydrochloride
Number analyzed (Participants) | 170
Age, Continuous [Mean (Standard Deviation); unit: Years] | 74.82 (7.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 123
  Male | 47

OUTCOME MEASURES:

1. Primary Outcome: Overall Summary of Adverse Events (AEs)
Description: Safety of study drug was assessed by clinical laboratory assessments, vital signs, weight, 12-lead electrocardiogram (ECG), physical and neurological examination. Treatment-Emergent Adverse Events (TEAEs) were defined as any event not present prior to the initiation of study treatment or any event already present that worsens in either intensity or frequency following exposure to study treatment. Serious adverse events were defined as AEs that led to or were life-threatening, resulted in or prolonged hospitalization, caused important or long-lasting disability, caused congenital abnormality or malformation, or resulted in death. Adverse drug reactions were defined as any harmful or unintended reaction to study treatment and were considered possibly related or probably related to study drug. Specific AEs and SAEs due to changes in clinical laboratory assessments, vital signs, weight, ECG, and physical and neurological exam are listed in the safety section.
Time Frame: Baseline (Day 1) up to Week 24
Population: as for baseline characteristics
Measure: Number; unit: Percentage of participants
Arm/Group | Donepezil Hydrochloride
Number analyzed (Participants) | 170
Percentage of participants
  AEs | 67.65
  ADRs | 47.06
  SAEs | 7.06
  Serious ADRs | 0.59

2. Secondary Outcome: Change From Baseline in the Mini-Mental State Examination (MMSE) Score
Description: The MMSE was used to measure cognitive impairment. The MMSE can evaluate overall cognitive function, and is widely used for the assessment of cognitive impairment in dementia patients. The questionnaire consists of 11 items, and each item aims to evaluate different cognitive domains such as orientation, memory, attention, and construction. The score ranged from 0 to 30, with a higher score indicating better function. A positive change score indicated improvement from baseline. The mean change was analyzed by Wilcoxon's signed rank test.
Time Frame: Baseline, Week 12, and Week 24 (Final visit)
Population: Efficacy analysis population included all participants who took at least one dose of study drug and had at least one baseline and at least one post-baseline assessment of the efficacy parameter. Twenty participants had no efficacy variables collected.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Donepezil Hydrochloride
Number analyzed (Participants) | 150
Scores on a scale
  Change W12 | -0.31 (2.76)
  Change W24 | -0.40 (2.75)

3. Secondary Outcome: Change From Baseline in the Neuropsychiatric Inventory Questionnaire (NPI-Q) Severity and Distress Total Scores
Description: The NPI-Q assessed twelve behavioral domains common in dementia including; hallucinations, delusions, agitation/aggression, dysphoria/depression, anxiety, irritability, disinhibition, euphoria, apathy, aberrant motor behavior, sleep/night-time behavior change, and appetite/eating change. The questionnaire is given by the clinician to the patient's caregiver who was asked if the behavior described is present in the patient. If "Yes", the informant then rates both the Severity of the symptoms present within the last month on a 3-point scale (1 = mild, 2= moderate, and 3= severe) and the associated impact of the symptom manifestations on them (i.e. Caregiver Distress) using a 5-point scale (0 = not distressing at all, 1 = minimal, 2 = mild, 3 = moderate, 4 = severe, and 5 = extreme or very severe). The total severity score represents the sum of individual scores and ranges from 0 to 36. The total distress score represents the sum of individual symptom scores and ranges from 0 to 60.
Time Frame: Baseline, Week 12, and Week 24 (Follow up visit)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Donepezil Hydrochloride
Number analyzed (Participants) | 150
Scores on a scale
  Change Week 12 (Severity) | 0.33 (4.74)
  Change Week 24 (Severity) | 0.09 (5.67)
  Change Week 12 (Distress) | 0.19 (6.83)
  Change Week 24 (Distress) | 0.29 (7.60)

ADVERSE EVENTS:
Time Frame: AEs were collected from Day 1 through Week 24 of study.
Description: Safety population included all participants who received at least one dose of study treatment and had at least one postbaseline safety assessment. Summary and analysis of adverse events were analyzed using TEAEs.
Arm/Group | Donepezil Hydrochloride
Serious Adverse Events (participants affected / at risk) | 12/170
Other Adverse Events (participants affected / at risk) | 109/170
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Donepezil Hydrochloride (N=170)
Femur fracture (Injury, poisoning and procedural complications) | 2
Rib fracture (Injury, poisoning and procedural complications) | 2
Ankle fracture (Injury, poisoning and procedural complications) | 1
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1
Ligament injury (Injury, poisoning and procedural complications) | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Gait disturbance (General disorders) | 1
Pneumonia (Infections and infestations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Donepezil Hydrochloride (N=170)
Nausea (Gastrointestinal disorders) | 21
Vomiting (Gastrointestinal disorders) | 19
Diarrhoea (Gastrointestinal disorders) | 11
Dizziness (Nervous system disorders) | 13
Lethargy (Nervous system disorders) | 8
Decreased appetite (Metabolism and nutrition disorders) | 16
Dyspepsia (Gastrointestinal disorders) | 5
Headache (Nervous system disorders) | 6
Somnolence (Nervous system disorders) | 6
Abdominal discomfort (Gastrointestinal disorders) | 2
Gastrointestinal disorder (Gastrointestinal disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 2
Faecal incontinence (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 1
Dental caries (Gastrointestinal disorders) | 1
Sedation (Nervous system disorders) | 2
Tremor (Nervous system disorders) | 2
Dreamy state (Nervous system disorders) | 1
Drooling (Nervous system disorders) | 1
Dysarthria (Nervous system disorders) | 1
Facial spasm (Nervous system disorders) | 1
Hypersomnia (Nervous system disorders) | 1
Paraesthesia (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 6
Insomnia (Psychiatric disorders) | 5
Aggression (Psychiatric disorders) | 4
Behavioural and psychiatric symptoms of dementia (Psychiatric disorders) | 3
Depression (Psychiatric disorders) | 3
Irritability (Psychiatric disorders) | 2
Sleep disorder (Psychiatric disorders) | 2
Compulsions (Psychiatric disorders) | 1
Compulsive hoarding (Psychiatric disorders) | 1
Confusional state (Psychiatric disorders) | 1
Delusion (Psychiatric disorders) | 1
Depressed mood (Psychiatric disorders) | 1
Disinhibition (Psychiatric disorders) | 1
Nightmare (Psychiatric disorders) | 1
Restlessness (Psychiatric disorders) | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 2
Hypophagia (Metabolism and nutrition disorders) | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Electrocardiogram QT prolonged (Investigations) | 5
Weight decreased (Investigations) | 5
Blood glucose increased (Investigations) | 2
Glucose urine present (Investigations) | 2
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Blood cholesterol increased (Investigations) | 1
Blood creatine phosphokinase increased (Investigations) | 1
Blood triglycerides increased (Investigations) | 1
Electrocardiogram ST segment elevation (Investigations) | 1
Electrocardiogram T wave abnormal (Investigations) | 1
Asthenia (General disorders) | 4
Fatigue (General disorders) | 3
Gait disturbance (General disorders) | 1
Chills (General disorders) | 1
Oedema (General disorders) | 1
Pain (General disorders) | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1
Contusion (Injury, poisoning and procedural complications) | 2
Urinary incontinence (Renal and urinary disorders) | 6
Acute kidney injury (Renal and urinary disorders) | 1
Enuresis (Renal and urinary disorders) | 1
Incontinence (Renal and urinary disorders) | 1
Nocturia (Renal and urinary disorders) | 1
Pollakiuria (Renal and urinary disorders) | 1
Nasopharyngitis (Infections and infestations) | 1
Periodontitis (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2
Cold sweat (Skin and subcutaneous tissue disorders) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1
Atrioventricular block second degree (Cardiac disorders) | 2
Bradycardia (Cardiac disorders) | 1
Hypertension (Vascular disorders) | 2
Pallor (Vascular disorders) | 1
Eye pain (Eye disorders) | 1
Hypersensitivity (Immune system disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other